CLINICAL TRIAL: NCT00282672
Title: Ablation of Intestinal Metaplasia Containing Dysplasia (AIM Dysplasia Trial) A Multi-center, Randomized, Sham-Controlled Trial: Protocol Amendment to Extend Follow-up to 5 Years
Brief Title: Ablation of Intestinal Metaplasia Containing Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B-204
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Barrett Esophagus
Keywords: Barrett's Esophagus; Dysplasia; Radiofrequency Ablation
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LGD Sham Procedure first then LGD Radiofrequency Ablation (Sham Comparator): Sham procedure plus anti-secretory medication. Subjects with Low Grade Dysplasia (LGD) receive proton pump inhibitor (PPI) with dose of Esomeprazole 40 mg BID.
  At 12 month, subjects crossover to receive radiofrequency ablation.
  Interventions: Device: Sham procedure plus anti-secretory medication
- LGD:Radiofrequency ablation (Active Comparator): Ablation System plus anti-secretory medication. Subjects with Low Grade Dysplasia (LGD) undergo an upper endoscopy with sizing of the esophageal diameter followed by radiofrequency ablation plus standard anti-secretory therapy (proton pump inhibitor, PPI-dose: Esomeprazole 40 mg BID.)
  Interventions: Device: Ablation System plus anti-secretory medication
- HGD Sham Procedure first then HGD Radiofrequency Ablation (Sham Comparator): Sham procedure plus anti-secretory medication. Subjects with High Grade Dysplasia (HGD) with proton pump inhibitor (PPI) dose: Esomeprazole 40 mg BID.
  At 12 month, subjects crossover to receive radiofrequency ablation.
  Interventions: Device: Sham procedure plus anti-secretory medication
- HGD:Radiofrequency ablation (Active Comparator): Ablation System plus anti-secretory medication. Subjects with High Grade Dysplasia (HGD) undergo an upper endoscopy with sizing of the esophageal diameter followed by radiofrequency ablation plus standard anti-secretory therapy (proton pump inhibitor, PPI-dose: Esomeprazole 40 mg BID.)
  Interventions: Device: Ablation System plus anti-secretory medication

INTERVENTIONS:
Device: Ablation System plus anti-secretory medication — Treatment group subjects undergo up to 4 ablation procedures (circumferential or focal) plus standard anti-secretory drug therapy (proton pump inhibitor, PPI).
  Other Names: HALO 360; HALO 90
  Arms: HGD:Radiofrequency ablation; LGD:Radiofrequency ablation
Device: Sham procedure plus anti-secretory medication — The Sham Control group undergo an upper endoscopy procedure with sizing of the esophageal diameter (a component of the ablation procedure steps, deemed the sham procedure) plus standard anti-secretory drug therapy (Proton pump inhibitor, PPI)
  Arms: HGD Sham Procedure first then HGD Radiofrequency Ablation; LGD Sham Procedure first then LGD Radiofrequency Ablation

SUMMARY:
The purpose of this study is to determine if the intervention of a 510(k)-cleared endoscopically-guided (Halo Ablation systems), ablation system plus anti-secretory therapy is better than anti-secretory therapy alone in clearing Barrett's Esophagus.

DETAILED DESCRIPTION:
Barrett's esophagus or intestinal metaplasia (IM) is a change in the epithelial lining of the esophagus. Barrett's esophagus develops as a result of chronic exposure of the esophagus to refluxed stomach acid and enzymes, as well as bile, resulting in recurrent mucosal injury. Injury is accompanied by inflammation and, ultimately, a cellular change (metaplasia) to a specialized columnar epithelium (Spechler SJ. Barrett's Esophagus. N Engl J Med 2002;346(11):836-842.)

Patients who have a diagnosis of Barrett's esophagus typically undergo surveillance endoscopy every 1-3 years with multiple biopsy specimens obtained to facilitate early detection of progression of IM to dysplasia (more severe precancerous changes) and adenocarcinoma. (Sampliner RE. Updated guidelines for the diagnosis, surveillance, and therapy of Barrett's esophagus. Am J Gastro 2002;97:1888-1895.) Progression of IM to low-grade dysplasia (LGD) indicates that cells exhibit more "cancer-like" architecture, thus warranting an accelerated surveillance endoscopy and biopsy program every 6 months rather than every 1-3 years as indicated for non-dysplastic IM. Progression to high-grade dysplasia (HGD) indicates that the cells are even more "cancer-like", thus warranting an even higher frequency surveillance endoscopy and biopsy program (every 3 months). Many HGD patients may undergo photodynamic therapy (PDT) or surgical esophagectomy, rather than remain in a frequent surveillance program. This more aggressive therapy is warranted because of the high rate of progression of HGD to adenocarcinoma.

Esophageal adenocarcinoma most commonly occurs after an insidious progression from IM to LGD to HGD. Therefore, surveillance is increased upon diagnosis of worsening grades of dysplasia. The incidence of esophageal adenocarcinoma is rapidly increasing as middle-aged and elderly demographic sub-groups expand (Peters JH, Hagen JA, DeMeester SR. Barrett's Esophagus. J Gastrointest Surg 2004;8(1):1-17.) In 2004, the American Cancer Society reported that there were 14,250 new cases of esophageal cancer, and 13,300 deaths attributable to esophageal cancer (www.cancer.org). The U.S. National Cancer Institute Surveillance, Epidemiology and End Results Program reported that the increasing incidence of esophageal adenocarcinoma was greater than for any other cancer in the United States (www.cancer.gov).

Elimination of the diseased epithelium containing IM with dysplasia is an intuitively favorable step for patients with this diagnosis. In other disease states, such as colon polyps or premalignant skin lesions, removal of the premalignant tissue results in a reduction in the risk of ultimately developing cancer. This is a logical conclusion when considering the premalignant lesion of Barrett's esophagus (particularly Barrett's esophagus with dysplasia), as the "tissue at risk" can be completely removed by ablation. This premise has been tested in the Barrett's dysplasia population in photoablative trials using PDT for patients with HGD, where PDT imparted a 50% reduction in risk over controls for the development of adenocarcinoma (Overholt BF, Panjehpour M, Haydek JM. Photodynamic therapy for Barrett's esophagus: follow-up. Gastrointest Endosc 1999;49(1):1-7.) The AIM Dysplasia Trial primary endpoints are removal of all dysplasia and IM, rather than detection of a difference in progression to adenocarcinoma or higher grades of dysplasia.

ELIGIBILITY:
Inclusion Criteria:1.Subject is 18-80 years of age, inclusive. 2.Subject has documented diagnosis of IM, maximum endoscopic length of 8 cm (as measured endoscopically from the TGF to the most proximal extent of the IM; i.e. TGF-TIM containing dysplasia as follows:

1. For LGD:i.LGD documented on biopsy within previous 12 months from enrollment while subject on PPI therapy.

   ii.Histology slides reviewed at central pathology service for trial confirm LGD on first confirmatory central pathology review or, if necessary, confirm LGD on a tie-breaker review by a second pathologist.
2. For HGD:i.Regular, non-nodular, non-ulcerated mucosa. ii.HGD documented on biopsy within previous 6 months from enrollment. iii.Histology slides reviewed at central pathology service for Trial confirm HGD on first confirmatory review or, if necessary, confirm HGD on a tie-breaker review by a second pathologist.

   iv.Baseline EUS within previous 12 months; 1.Catheter-based EUS excludes suspicious thickened Barrett's areas or, if suspicious areas found, prompts stacked biopsies of thickened area, the results of which do not render subject ineligible for enrollment.

   3.For subjects with EMR history,the documented diagnosis of IM with dysplasia meets criterion #2 from biopsies collected either after the EMR procedure or during the EMR procedure but not from the EMR site.

   4.Subject able to take oral proton pump inhibitor medication. 5.Subject able to discontinue aspirin and/or non-steroidal anti-inflammatory medications 7 days before and after all ablation procedures.

   6.For female subjects of childbearing potential, a negative pregnancy test within 2 weeks of randomization.

   7.Subject eligible for treatment and follow-up endoscopy and biopsy as required by the Protocol.

   8.Subject willing to provide written, informed consent to participate in this clinical study and understands the responsibilities of trial participation.

   Exclusion Criteria:1.The subject is pregnant or planning a pregnancy during the study period.

   2.Esophageal stricture preventing passage of endoscope or catheter. 3.Active esophagitis described as erosions or ulcerations encompassing more than 10% of distal esophagus.

   4.Any history of malignancy of the esophagus. 5.Prior radiation therapy to the esophagus,except head and neck region radiation therapy.

   6.Any previous ablative therapy within the esophagus (PDT, MPEC, APC, laser treatment, other).

   7.History of EMR that meets any of the following criteria:a.EMR performed less than 8 weeks prior to the randomization endoscopy encounter

b.EMR performed in a wide field manner (encompassing more than 90 degrees of any area of the esophagus.

8.Any previous esophageal surgery, including except fundoplication without complications (i.e. no slippage, dysphagia, etc).

9.Evidence of esophageal varices during treatment endoscopy. 10.Report of uncontrolled coagulopathy with international normalized ratio (INR) > 1.3 or platelet count <75,000 platelets per µL 11.Subject has a life-expectancy of less than two years due to an underlying medical condition.

12.Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.

13.Subject has an implantable pacing device (examples; AICD, neurostimulator, cardiac pacemaker)and has not received clearance for enrollment in this study by specialist responsible for the pacing device.

14.The subject is currently enrolled in an investigational drug or device trial that clinically interferes with the AIM Dysplasia Trial endpoints.

15.Subject suffers from psychiatric or other illness deemed by the investigator as an inability to comply with protocol.

For the 5 year extension, patient must have:1. Enrolled in the B-204 protocol. 2. Completed 1 year follow-up. 3. Completed 2 year follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-02; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (19):
- United States (19):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arizona, VAMC, Tucson, Arizona
  - UC Irvine Medical Center, Orange, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Harvard, VA Boston Healthcare W Roxbury, West Roxbury, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Kansas School of Medicine - Veterans Affairs Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - UNC Center for Functional GI & Motility Disorders, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastrointestinal Associates, Knoxville, Tennessee
  - VAMC Dallas, Dallas, Texas
  - Tacoma Digestive Disease Research Center, Tacoma, Washington

REFERENCES:
- [Background] Dunkin BJ, Martinez J, Bejarano PA, Smith CD, Chang K, Livingstone AS, Melvin WS. Thin-layer ablation of human esophageal epithelium using a bipolar radiofrequency balloon device. Surg Endosc. 2006 Jan;20(1):125-30. doi: 10.1007/s00464-005-8279-9. Epub 2005 Dec 7. PMID 16333533
- [Background] Ganz RA, Utley DS, Stern RA, Jackson J, Batts KP, Termin P. Complete ablation of esophageal epithelium with a balloon-based bipolar electrode: a phased evaluation in the porcine and in the human esophagus. Gastrointest Endosc. 2004 Dec;60(6):1002-10. doi: 10.1016/s0016-5107(04)02220-5. PMID 15605025
- [Result] Shaheen NJ, Sharma P, Overholt BF, Wolfsen HC, Sampliner RE, Wang KK, Galanko JA, Bronner MP, Goldblum JR, Bennett AE, Jobe BA, Eisen GM, Fennerty MB, Hunter JG, Fleischer DE, Sharma VK, Hawes RH, Hoffman BJ, Rothstein RI, Gordon SR, Mashimo H, Chang KJ, Muthusamy VR, Edmundowicz SA, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Falk GW, Kimmey MB, Madanick RD, Chak A, Lightdale CJ. Radiofrequency ablation in Barrett's esophagus with dysplasia. N Engl J Med. 2009 May 28;360(22):2277-88. doi: 10.1056/NEJMoa0808145. PMID 19474425
- [Result] Shaheen NJ, Overholt BF, Sampliner RE, Wolfsen HC, Wang KK, Fleischer DE, Sharma VK, Eisen GM, Fennerty MB, Hunter JG, Bronner MP, Goldblum JR, Bennett AE, Mashimo H, Rothstein RI, Gordon SR, Edmundowicz SA, Madanick RD, Peery AF, Muthusamy VR, Chang KJ, Kimmey MB, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Dumot JA, Falk GW, Galanko JA, Jobe BA, Hawes RH, Hoffman BJ, Sharma P, Chak A, Lightdale CJ. Durability of radiofrequency ablation in Barrett's esophagus with dysplasia. Gastroenterology. 2011 Aug;141(2):460-8. doi: 10.1053/j.gastro.2011.04.061. Epub 2011 May 6. PMID 21679712
- [Derived] Shaheen NJ, Peery AF, Overholt BF, Lightdale CJ, Chak A, Wang KK, Hawes RH, Fleischer DE, Goldblum JR; AIM Dysplasia Investigators. Biopsy depth after radiofrequency ablation of dysplastic Barrett's esophagus. Gastrointest Endosc. 2010 Sep;72(3):490-496.e1. doi: 10.1016/j.gie.2010.04.010. Epub 2010 Jul 3. PMID 20598302

RESULTS

PARTICIPANT FLOW:
Groups:
- LGD Sham Procedure First Then LGD Radiofrequency Ablation; HGD Sham Procedure First Then HGD Radiofrequency Ablation: After the 1 year follow up was completed, all sham patients were offered cross-over to receive RFA.
Period: 1 Year
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Started | 22 | 42 | 21 | 42
Completed | 19 | 40 | 20 | 38
Not Completed | 3 | 2 | 1 | 4
Period: 2 Year: Sham Crossed Over to RFA
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Started | 19 (19 crossed over to RFA treatment) | 40 | 16 (16 Crossed over to RFA treatment) | 38
Completed | 16 | 39 | 15 | 36
Not Completed | 3 | 1 | 1 | 2
Period: 5 Year: Follow up
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Started | 15 (1 withdrew) | 32 (7 withdrew) | 12 (3 withdrew) | 25 (11 withdrew)
Completed | 14 | 27 | 12 | 20
Not Completed | 1 | 5 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- HGD Sham Procedure First Then LGD Radiofrequency Ablation: After the 1 year follow up was completed, all sham patients were offered cross-over to receive RFA.
- Total: Total of all reporting groups
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then LGD Radiofrequency Ablation | HGD Radiofrequency Ablation | Total
Number analyzed (Participants) | 22 | 42 | 21 | 42 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (1.9) | 66.3 (1.4) | 67.3 (1.8) | 65.9 (1.4) | 65.95 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 0 | 5 | 17
  Male | 19 | 33 | 21 | 37 | 110
Region of Enrollment [Number; unit: participants]
  United States | 22 | 42 | 21 | 42 | 127

OUTCOME MEASURES:

1. Primary Outcome: The % of Patients With Complete Eradication of Intestinal Metaplasia (IM) at 12 Month
Description: % of patients with complete eradication of IM out of the number of participants analyzed at 12 month was calculated.
Time Frame: 12 month
Population: LGD: Radiofrequency group- 2 patients withdrew and were not analyzed, HGD: Radiofrequency Ablation: 4 patients withdrew and were not analyzed. LGD Sham procedure first then LGD Radiofrequency Ablation group and HGD Sham procedure first then HGD Radiofrequency Ablation group were not analyzed to measure the CR-IM at one year.
Measure: Number; unit: percentage of participants
Arm/Group | LGD:Radiofrequency Ablation | HGD:Radiofrequency Ablation
Number analyzed (Participants) | 40 | 38
percentage of participants | 85 | 81.5

2. Primary Outcome: The % of Patients With Complete Eradication of Dysplasia at 12 Month
Description: % of patients with complete eradication of Dysplasia out of the number of participants analyzed at 12 month was calculated.
Time Frame: 12 month
Population: LGD: Radiofrequency group- 2 patients withdrew and were not analyzed, HGD: Radiofrequency Ablation: 4 patients withdrew and were not analyzed. LGD Sham procedure first then LGD Radiofrequency Ablation group and HGD Sham procedure first then HGD Radiofrequency Ablation group were not analyzed to measure the CR-D at one year.
Measure: Number; unit: percentage of participants
Arm/Group | LGD:Radiofrequency | HGD:Radiofrequency
Number analyzed (Participants) | 40 | 38
percentage of participants | 95 | 89.5

3. Primary Outcome: The % of Patients With Complete Histological Clearance of Intestinal Metaplasia at 24 Months.
Description: % of patients with complete eradication of IM out of the number of participants analyzed at 24 month was calculated.
Time Frame: 24 Month
Measure: Number; unit: percentage of participants
Groups:
- LGD Sham Procedure First Then LGD Radiofrequency Ablation: Crossed over to LGD:Radiofrequency
- HGD Sham Procedure First Then HGD Radiofrequency Ablation: Crossed over to HGD: Radiofrequency
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD:Radiofrequency | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Number analyzed (Participants) | 16 | 39 | 15 | 36
percentage of participants | 100 | 97.4 | 93.3 | 88.9

4. Primary Outcome: 5 Year Extension: % of All Patients Enrolled in the Extension Protocol and Available for Analysis Demonstrating CR-IM at 5 Years
Description: For patient who made it to the 5 year visit, % of patients demonstrating complete eradication of intestinal metaplasia (CE-IM) was calculated.
Time Frame: 5 years
Population: patient who made it to the 5 year visit
Measure: Number; unit: percentage of participants
Groups:
- All LGD Patients: LGD: Sham procedure group crossed over to LGD: Radiofrequency group at 12 month
- All HGD Patients: HGD: Sham procedure group crossed over to HGD: Radiofrequency group at 12 month
Arm/Group | All LGD Patients | All HGD Patients
Number analyzed (Participants) | 41 | 32
percentage of participants | 85.3 | 96.8

5. Primary Outcome: Durability of Eradication With no Additional Treatments
Time Frame: 5 year
Population: 41 LGD subjects and 32 HGD subjects completed 5 year visit
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 73
percentage of participants | 75

6. Primary Outcome: 5 Year Extension: % of All Patients Enrolled in the Extension Protocol and Available for Analysis Demonstrating CR-D at 5 Years
Description: For patient who made it to the 5 year visit, % of patients demonstrating complete eradication of dysplasia was calculated and all were free of dysplasia
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | All LGD Patients | All HGD Patients
Number analyzed (Participants) | 41 | 32
percentage of participants | 100 | 96.8

7. Secondary Outcome: The % of Patients With Complete Histological Clearance of IM at 12 Months, Comparing Treatment Versus Sham Control Groups Within a Specific Dysplasia Subgroup
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | LGD Radiofrequency Ablation | LGD Sham Procedure First Then LGD Radiofrequency Ablation | HGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation
Number analyzed (Participants) | 40 | 18 | 38 | 15
percentage of participants | 85 | 72.2 | 81.5 | 80

8. Secondary Outcome: Within the HGD Subgroup, the % of Patients With Complete Histological Clearance of HGD (CR-D) at 12 Months, Comparing Treatment Versus Sham Control Groups.
Time Frame: 12 Month
Population: 16 HGD Sham procedure subjects crossed over to RFA treatment after one year
Measure: Number; unit: percentage of participants
Arm/Group | HGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation
Number analyzed (Participants) | 38 | 15
percentage of participants | 89.4 | 86.6

9. Secondary Outcome: Histological Clearance of IM (% Biopsies)
Description: % of patients with histological clearance of IM out of the number of participants analyzed at 12 month was calculated.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | LGD Radiofrequency Ablation | LGD Sham Procedure First Then LGD Radiofrequency Ablation | HGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation
Number analyzed (Participants) | 40 | 18 | 38 | 15
percentage of participants | 85 | 72.2 | 81.5 | 80

10. Secondary Outcome: Progression of Dysplasia (i.e., HGD to Adenocarcinoma, or LGD to HGD or Adenocarcinoma)
Time Frame: 5 year
Measure: Number; unit: participants
Arm/Group | LGD to HGD | LGD to IMC | HGD to IMC
Number analyzed (Participants) | 47 | 47 | 37
participants | 5 | 1 | 1

11. Secondary Outcome: Subject Discomfort : Chest Pain Score on Day 1
Description: Chest pain score was measured on a visual analogue scale of 0 to 100, with higher scores indicating a greater severity of pain
Time Frame: Day 1 , if ablated
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Number analyzed (Participants) | 20 | 40 | 20 | 41
Scores on a scale | 0 [0 to 0] | 26 [4 to 48] | 0 [0 to 0] | 22 [0 to 57]

12. Secondary Outcome: Quality of Life Questionnaire (Baseline v. 12 and 24 Mos)
Time Frame: 0, 12, and 24 months
Population: Data had not been collected consistently to analyze the data.
Arm/Group | All Groups
Number analyzed (Participants) | 0

13. Secondary Outcome: Adverse Event Incidence
Description: Data reported in the adverse event section
Time Frame: 12 months for Treatment and Sham Comparison
Measure: Number; unit: Adverse event occurrences
Groups:
- Sham Patients: Patients randomized to Sham Procedure arm.
- Treatment Patients: Patients randomized to Radiofrequency Ablation at start of study and underwent RFA treatment at randomization.
Arm/Group | Sham Patients | Treatment Patients
Number analyzed (Participants) | 43 | 84
Adverse event occurrences
  AE's related to procedure | 7 | 32
  AE's unrelated to procedure | 17 | 34

14. Secondary Outcome: For 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension and Available for Analysis at 5 Years Demonstrating Any Adenocarcinoma in Any Biopsy Obtained From the Esophageal Body Since Primary RFA (0-5 Years)
Time Frame: 5 years
Population: 41 LGD patients and 21 HGD subjects completed the 5 year study and used for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 73
percentage of participants | 2.7

15. Secondary Outcome: 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension and Available for Analysis at 5 Years Demonstrating Any Adenocarcinoma in Any Biopsy Obtained From the Esophageal Body After 2 Years and Inclusive of the 5 Year Visit
Time Frame: 5 years
Population: Similar analysis was performed and the result is provided for the outcome measure #14. The data were collected to answer the outcome measure #14.
Arm/Group | All Groups
Number analyzed (Participants) | 0

16. Secondary Outcome: 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension Protocol and Available for Analysis Demonstrating CR-IM at 5 Year
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 41
percentage of participants | 85.4

17. Secondary Outcome: 5 Year Extension:Proportion (%) of All Patients Enrolled in This Extension Protocol and Available for Analysis Demonstrating CR-D at 5 Year
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 41
percentage of participants | 100

18. Secondary Outcome: 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension Protocol and Available for Analysis Demonstrating CR-IM at 4 Year
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 43
percentage of participants | 79.1

19. Secondary Outcome: 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension Protocol and Available for Analysis Demonstrating CR-IM at 3 Year
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 42
percentage of participants | 92.9

20. Secondary Outcome: 5 Year Extension: Proportion (%) of All Patients Enrolled in This Extension Protocol and Available for Analysis Demonstrating CR-D at 4 Year
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 43
percentage of participants | 93

21. Secondary Outcome: 5 Year Extension: Serious Adverse Event Incidence
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 127
participants
  Bleed | 1
  Chest Pain | 3

22. Secondary Outcome: 5 Year Extension: All Cause Mortality of the Group From 2 to 5 Years.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | All Groups
Number analyzed (Participants) | 127
percentage of participants | 0

ADVERSE EVENTS:
Arm/Group | LGD Sham Procedure First Then LGD Radiofrequency Ablation | LGD Radiofrequency Ablation | HGD Sham Procedure First Then HGD Radiofrequency Ablation | HGD Radiofrequency Ablation
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/42 | 0/21 | 2/42
Other Adverse Events (participants affected / at risk) | 4/22 | 11/42 | 7/21 | 12/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGD Sham Procedure First Then LGD Radiofrequency Ablation (N=22) | LGD Radiofrequency Ablation (N=42) | HGD Sham Procedure First Then HGD Radiofrequency Ablation (N=21) | HGD Radiofrequency Ablation (N=42)
PAIN, NAUSEA, VOMITTING, FULLNESS, ABDOMINAL DISCOMFORT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper GI Bleed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGD Sham Procedure First Then LGD Radiofrequency Ablation (N=22) | LGD Radiofrequency Ablation (N=42) | HGD Sham Procedure First Then HGD Radiofrequency Ablation (N=21) | HGD Radiofrequency Ablation (N=42)
MUCOSAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
MELENA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STRICTURE REQUIRING DILATATION (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 2 (3) | 4 (4)
VOMITTING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
CHEST PAIN/ THROAT PAIN / NAUSEA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
STRICTURE / SCARRING (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
BLOATED, REFLUX SENSATION, DIFFICULTY SWALLOWING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NARROWED ESOPHAGUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESOPHAGEAL VARICES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEVER; DIARRHEA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAINFUL SWALLOWING / CHEST PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
PREMATURE FULLNESS WITH MEALS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAINFUL SWALLOWING, ABDOMINAL PAIN, CHEST PAIN. (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEVER, LARYNGITIS, PHARYNGITIS AND BRONCHITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEVERE NAUSEA,VOMITING, ULCERATION, WEIGHT LOSS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ULCERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
EROSIVE ESOPHAGEAL MUCOSA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIGHT EAR ACHE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
PAIN; ELEVATED BP (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less